CLINICAL TRIAL: NCT02480998
Title: A Randomized, Double-blind, Active Comparator, Phase I/Ⅱa Clinical Trial to Assess the Safety and Immunogenicity of the 'IL-YANG Flu Vaccine Quadrivalent Inj.' in Healthy Korean Adult Subjects
Brief Title: Study to Evaluate the Safety and Immunogenicity of 'IL-YANG Flu Vaccine Quadrivalent Inj' in Healthy Korean Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IY_IFEZ_Q120
Record Dates: First submitted 2015-06-11; First posted 2015-06-25 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IL-YANG Flu Vaccine QIV 0.5mL (Experimental): A single 0.5mL dose administrated as an intramuscular injection.
  Interventions: Biological: IL-YANG Flu Vaccine QIV 0.5mL
- IL-YANG Flu Vaccine TIV 0.5mL (Active Comparator): A single 0.5mL dose administrated as an intramuscular injection.
  Interventions: Biological: IL-YANG Flu Vaccine TIV 0.5mL

INTERVENTIONS:
Biological: IL-YANG Flu Vaccine QIV 0.5mL
  Arms: IL-YANG Flu Vaccine QIV 0.5mL
Biological: IL-YANG Flu Vaccine TIV 0.5mL
  Arms: IL-YANG Flu Vaccine TIV 0.5mL

SUMMARY:
This study evaluates the safety, tolerability and immunogenicity of IL-YANG quadrivalent vaccine versus IL-YANG trivalent vaccine after a single intramuscular administration in healthy Korean males and females 19 to < 65 years of age.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, phase I/Ⅱa clinical trial.

During the Part A phase, all safety data collected from the 12 subjects enrolled in the Part A phase will be analyzed to determine the safety and tolerability of the investigational product, which should include any solicited and unsolicited adverse drug reactions occurring for the first 7 days after vaccination and any adverse events occurring for 28 days after vaccination. Antibody titer test will be also performed to evaluate the efficacy (immunogenicity) of the investigational product. During the Part B phase, a total of 72 subjects will be enrolled, and all safety data (including all adverse events) and immunogenicity data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women 19 to < 65 years of age at screening
* Body weight within ±20% of ideal body weight at screening
* Women of childbearing potential must have a negative serum beta-hCG at visit 2; and agree to use a proper contraceptive method for 1 month after vaccination (starting from 3 months before screening), using a medication or device that does not have any drug-interaction with the investigational product.
* Subjects with no congenital or chronic disease who were considered suitable for the study after screening assessments (investigator's opinion, medical history, physical examination, laboratory test, chest X-ray, and ECG) conducted no later than 28 days prior to vaccination
* Subjects who were given, and fully understood, the information about the study, and have provided voluntary written informed consent to participate in the study and to comply with all applicable study requirements

Exclusion Criteria:

* Subject with known allergy to eggs, chicken, or any components of the investigational product
* Subjects who had received an influenza vaccine within the last 6 months prior to study entry
* Subjects who have known or suspected infection with HAV, HBV, HCV, HIV or VDRL
* Subjects who have concurrent or a past history of, immune deficiency disease
* Subject with a history of Guillain-Barre syndrome
* Subject with hemophilia or thrombocytopenia or being treated with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection
* Subjects with known allergy to a drug, food or latex, who had a history of anaphylaxis
* Subjects who had an acute fever with body temperature > 38.0 Cº within 72 hours prior to administration of the investigational product or symptoms of suspected acute disease within 14 days prior to administration of the investigational product
* Subjects who had received another vaccine within 28 days before administration of the investigational product or are planning to receive another vaccine during the study.
* Subjects who had participated in another clinical trial within the 30 days before administration of the investigational product.
* Subjects who had previously received blood-derived products (including immunoglobulin) within the last 3 months prior to administration of the Investigational product, or are scheduled to receive a treatment with blood-derived products during the study
* Subjects who had received, or are scheduled to receive, systemic immunosuppressive therapy, radiation therapy or high-dose steroid therapy within the last 6 months prior to administration of the study
* Subjects with a history of drug abuse within the last 6 months prior to vaccination, or is suspected of drug abuse
* Subjects with excessive consumption of caffeine, alcohol, or tobacco
* Subjects with other clinically significant medical or psychiatric illness who in the investigator's opinion, are not be suitable for the study

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IL-YANG Flu Vaccine QIV 0.5mL: A single 0.5mL dose administrated as an intramuscular injection.
  IL-YANG Flu Vaccine QIV 0.5mL
- IL-YANG Flu Vaccine TIV 0.5mL: A single 0.5mL dose administrated as an intramuscular injection.
  IL-YANG Flu Vaccine TIV 0.5mL
Period: Overall Study
Arm/Group | IL-YANG Flu Vaccine QIV 0.5mL | IL-YANG Flu Vaccine TIV 0.5mL
Started | 56 | 28
Completed | 56 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IL-YANG Flu Vaccine QIV 0.5mL | IL-YANG Flu Vaccine TIV 0.5mL | Total
Number analyzed (Participants) | 56 | 28 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.77 (7.01) | 27.75 (8.48) | 27.10 (7.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 45 | 23 | 68

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Rate
Description: Percentage of subjects achieving seroconversion* for HI antibody after vaccination
Time Frame: 28 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IL-YANG Flu Vaccine QIV 0.5mL | IL-YANG Flu Vaccine TIV 0.5mL
Number analyzed (Participants) | 56 | 28
percentage of participants
  H1N1 | 58.93 [46.04 to 71.81] | 64.29 [46.54 to 82.03]
  H3N2 | 64.29 [51.74 to 76.84] | 53.57 [35.10 to 72.04]
  B/Yamagata | 55.36 [42.34 to 68.38] | 35.71 [17.97 to 53.46]
  B/Victoria | 46.43 [33.37 to 59.49] | 14.29 [1.32 to 27.25]

2. Primary Outcome: Seroprotection Rate
Description: Percentage of subjects achieving seroprotection* for HI antibody after vaccination
Time Frame: 28 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IL-YANG Flu Vaccine QIV 0.5mL | IL-YANG Flu Vaccine TIV 0.5mL
Number analyzed (Participants) | 56 | 28
percentage of participants
  H1N1 | 94.64 [88.75 to 100.00] | 85.71 [72.75 to 98.68]
  H3N2 | 96.43 [91.57 to 100.00] | 82.14 [67.96 to 96.33]
  B/Yamagata | 87.50 [78.84 to 96.16] | 78.57 [63.37 to 93.77]
  B/Victoria | 78.57 [67.82 to 89.32] | 64.29 [46.54 to 82.03]

3. Secondary Outcome: GMR
Description: Geometric Mean Ratio of post vaccination HI geometric mean titers
Time Frame: 28 days
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of GMT titer
Groups:
- IL-YANG Flu Vaccine QIV 0.5mL: A single 0.5mL dose administrated as an intramuscular injection.
  IL-YANG Flu Vaccine QIV 0.5mL
  56
- IL-YANG Flu Vaccine TIV 0.5mL: A single 0.5mL dose administrated as an intramuscular injection.
  IL-YANG Flu Vaccine TIV 0.5mL
  28
Arm/Group | IL-YANG Flu Vaccine QIV 0.5mL | IL-YANG Flu Vaccine TIV 0.5mL
Number analyzed (Participants) | 56 | 28
Ratio of GMT titer
  H1N1 | 5.32 [3.39 to 8.35] | 8.41 [4.71 to 15.01]
  H3N2 | 6.90 [4.25 to 11.19] | 6.73 [3.411 to 14.57]
  B/Massachusetts | 3.85 [2.82 to 5.27] | 2.90 [1.67 to 5.03]
  B/Brisbane | 3.20 [2.52 to 4.06] | 2.00 [1.40 to 2.85]

4. Secondary Outcome: GMT
Description: Geometric Mean Titer of post vaccination HI geometric mean titers
Time Frame: 28 days
Measure: Geometric Mean (95% Confidence Interval); unit: HI titer of post vaccination
Arm/Group | IL-YANG Flu Vaccine QIV 0.5mL | IL-YANG Flu Vaccine TIV 0.5mL
Number analyzed (Participants) | 56 | 28
HI titer of post vaccination
  H1N1 | 128 [97.31 to 168.50] | 110.40 [69.30 to 175.80]
  H3N2 | 176.70 [132.10 to 234.20] | 128.00 [69.42 to 236.20]
  B/Massachusetts | 73.36 [58.97 to 91.27] | 51.24 [32.99 to 79.57]
  B/Brisbane | 52.52 [44.21 to 62.39] | 36.23 [28.51 to 46.03]

ADVERSE EVENTS:
Arm/Group | IL-YANG Flu Vaccine QIV 0.5mL | IL-YANG Flu Vaccine TIV 0.5mL
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/28
Other Adverse Events (participants affected / at risk) | 0/56 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes